CLINICAL TRIAL: NCT04231136
Title: An Open-label, Randomized, Crossover Study to Evaluate the Pharmacodynamics After Single Oral Dosing of Tegoprazan, EAPA115 and RAPA115 in Healthy Volunteers
Brief Title: Study to Evaluate the Pharmacodynamics After Single Oral Dosing of Tegoprazan, EAPA115 and RAPA115 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: HK inno.N Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CJ_APA_115
Record Dates: First submitted 2020-01-09; First posted 2020-01-18 (Actual); Last update posted 2020-12-01 (Actual); Status verified 2020-01

CONDITIONS: Healthy
MeSH Terms: interventions — tegoprazan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tegoprazan 50 mg (Experimental): Oral administration of Tegoprazan 50 mg tablet once a day
  Interventions: Drug: Tegoprazan 50 mg
- EAPA115 (Active Comparator): Oral administration of EAPA115 once a day
  Interventions: Drug: EAPA115
- RAPA115 (Active Comparator): Oral administration of RAPA115 once a day
  Interventions: Drug: RAPA115

INTERVENTIONS:
Drug: Tegoprazan 50 mg — Tegoprazan 50 mg tablet
  Other Names: K-CAB
  Arms: Tegoprazan 50 mg
Drug: EAPA115 — EAPA115
  Arms: EAPA115
Drug: RAPA115 — RAPA115
  Arms: RAPA115

SUMMARY:
This study aims to evaluate the pharmacodynamics after single oral dosing of tegoprazan, EAPA115 and RAPA115 in healthy volunteers.

DETAILED DESCRIPTION:
Evaluation Criteria

* Pharmacodynamic assessments with intragastric pH
* Safety assessments with adverse event monitoring including subjective/objective symptoms, physical examination, vital signs, electrocardiogram, and laboratory test

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 19 to 65 years (not inclusive) at the time of signing the informed consent form (ICF).
* Body mass index (BMI) ≥ 17.5 and < 30.5 kg/m^2 with a body weight ≥ 45 kg at screening. Body mass index (kg/m^2) = weight (kg)/height (m)^2
* Confirmed as H. pylori negative
* A subject without any congenital or chronic disease within 3 years, and has no medical examination result as pathological symptoms or signs.
* A subject determined eligible for this study based on the screening test such as clinical laboratory tests (hematology test, chemistry test, urine test, virus/bacteria test, etc.), vital signs, and electrocardiogram.
* A subject who is fully informed of the purpose and content of the study and agrees to participate in the study on its own will and signs the consent form approved by the Institutional Review Board (IRB) of the Seoul National University Hospital, prior to participate in the study.
* A subject who has the ability and willingness to participate throughout the whole study period.

Exclusion Criteria:

* A subject with clinically significant blood, renal, endocrine, respiratory, gastrointestinal, urinary, cardiovascular, hepatic, psychical, neurologic, or immunologic diseases (except for simple dental past history such as tartar, impacted tooth, or wisdom tooth) or evidence.
* A subject with a history of gastrointestinal disorders (esophageal diseases such as esophageal achalasia or esophageal stricture, Crohn's disease) or surgery (except for simple appendectomy, herniotomy, and tooth extraction surgery) that may affect the absorption of drugs.
* A subject with the *17 allele of CYP2C19 (Ultrarapid metabolizer).
* A subject with AST and ALT levels exceeding 3 times of the upper limit of the reference range in the screening test.
* A subject with a history of excessive caffeine (> 5 units/day) or regular alcohol consumption exceeding 210 g/week within 6 months of screening test. (1 glass of beer (5%) (250 mL) = 10 g, 1 shot of soju (20%) (50 mL) = 8 g, 1 glass of wine (12%) (125 mL) = 12 g)
* A subject who participated in other clinical trial or bioequivalence study and administered the study medication within 6 months prior to the first administration of the investigational product of this study.
* A subject with significant alcohol or drug abuse within a year of screening test.
* A subject who administered drugs that significantly induce or inhibit drug metabolizing enzymes within 30 days prior to the first administration of the investigational product of this study.
* A subject who smoked cigarettes more than 20 per day within 6 months of screening test.
* A subject who administered prescribed drug or over-the-counter drug within 10 days prior to the first administration of the investigational product of this study.
* A subject who has donated whole blood within 2 months or those who donated the component blood within 1 month prior to the first administration of the investigational product of this study.
* A subject who has hypersensitivity to the investigational product of this study, benzimidazoles, penicillin and macrolide and its related medical history.
* A subject with rare genetic problems such as fructose intolerance, glucose-galactose malabsorption, or sucrase-isomaltase deficiency.
* Pregnant or nursing women
* A subject who cannot use reliable contraception during the entire period of the clinical trial (e.g, condom use, intrauterine device, tubal ligation, cervical cap, contraceptive diaphragm, etc.).
* A subject who is judged by the investigator to be ineligible to participate in the test.

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2020-01-14 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-08-03 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic Evaluation | Pre-dose(0 hour) up to 24 hours after Investigational product administration in each period
  The ratio of duration(Duration %) with pH ≥ 4 over 24 hours
Pharmacodynamic Evaluation | Pre-dose(0 hour) up to 24 hours after Investigational product administration in each period
  The ratio of duration(Duration %) with pH ≥ 6 over 24 hours
Pharmacodynamic Evaluation | Pre-dose(0 hour) up to 24 hours after Investigational product administration in each period
  Median pH
Pharmacodynamic Evaluation | Pre-dose(0 hour) up to 24 hours after Investigational product administration in each period
  Mean pH
Pharmacodynamic Evaluation | Pre-dose(0 hour) up to 24 hours after Investigational product administration in each period
  Baseline pH and changes in pH after the administration of investigational products (change of duration %, change of mean pH, change of median pH)
Pharmacodynamic Evaluation | Pre-dose(0 hour) up to 12 hours after Investigational product administration in each period
  The ratio of duration(Duration %) with pH ≥ 4 during nocturnal period* (*12 hours after administration of investigational product)
Pharmacodynamic Evaluation | Pre-dose(0 hour) up to 12 hours after Investigational product administration in each period
  The ratio of duration(Duration %) with pH ≥ 6 during nocturnal period* (*12 hours after administration of investigational product)

CONTACTS AND LOCATIONS:
Overall Officials: In-Jin Jang, MD, PhD, Principal Investigator — Seoul National University Hospital, Dept. of Clinical Pharmacology
Locations (1):
- Seoul National University Hospital, Clinical Trial Center, Seoul, South Korea